CLINICAL TRIAL: NCT03109197
Title: The SUDC Registry and Research Collaborative
Brief Title: Sudden Unexplained Death in Childhood (SUDC) Registry
Acronym: SUDC
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Columbia University (Other); Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 14-01061
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Sudden Unexplained Death Syndrome; Sudden Unexplained Death in Childhood
MeSH Terms: conditions — Brugada Syndrome

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — For retrospective SUDC cases: Mucosal swab or blood samples for DNA analysis, pathology slides, tissue blocks, tissue samples or organs retained at autopsy.
  For prospective SUDC cases: Mucosal swab or blood samples for DNA analysis, pathology slides, tissue blocks, tissue samples except heart and brain tissue that will undergo full cardiac pathology consultation or neuropathology consultation will be transferred to pathologists at NYU or Mayo (based on pathologist availability).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective SUDC cases: All child biospecimens (including mucosal swab or blood samples for DNA analysis, pathology slides, tissue blocks, tissue samples or organs retained at autopsy) will be transferred to NYU Biorepository
  Interventions: Other: Biospecimin Collection
- Prospective SUDC cases: Heart and brain tissue will undergo full cardiac pathology consultation or neuropathology consultation will be transferred to pathologists at NYU or Mayo (based on pathologist availability). The PHI will remain intact in these cases since they will need to know how to identify the deceased with the medical records they receive and to complete the entire investigation thoroughly. A full consultation report will be sent back to Dr. Orrin Devinsky and tissue will be returned to the NYU biorepository upon completion of the cardiac or neuropathology consultation.
  Interventions: Other: Biospecimin Collection

INTERVENTIONS:
Other: Biospecimin Collection

SUMMARY:
The purpose is to increase the understanding of the characteristics, circumstances, medical histories and pathologies of children from ages 11 months through 18 years who have died suddenly and unexpectedly, and in some instances, without explanation. The SUDC Registry and Research Collaborative will analyze cases of sudden unexpected deaths in these children to understand risk factors and causes, and develop preventative measures.

DETAILED DESCRIPTION:
* Review the child's death, medical and family history by our study pathologists (including forensic, pediatric, cardiac and neuropathologists) to determine whether a possible, probable or definite cause of death can be identified and whether additional studies might be helpful in determining a specific cause of death.
* For case investigations that are open/active, the registry offers cardiac pathology, and neuroimaging/neuropathology consultations.
* For those cases determined to be unexplained/undetermined- access to genetic analysis (whole exome sequencing) when viable samples are available. Additional genetic analysis opportunities for biological parents and some family members. For more information, please see our Genetics Frequently Asked Questions.
* Study the risks that lead to sudden unexplained death in childhood (SUDC).
* Provide families with a review of their child's death through a case review report.
* Identify at-risk individuals with the hopes of gaining knowledge to establish prevention strategies to reduce the chances of sudden unexplained death in the future.

ELIGIBILITY:
Inclusion Criteria:

Retrospective SUDC Cases

* 11months to 18 years of age.
* Subjects whose cause of death was sudden and unexplained-"Postinfancy SIDS," "Sudden Death of Childhood," "Undetermined," "Late SIDS," a vague description of symptoms of "undetermined etiology," or a diagnosis acknowledged to be speculative by the prosecting pathologist
* If the retrospective case has banked DNA specimens.

Prospective SUDC Cases

* SUDC cases, parents and eligible family members from 11months-100 years of age.
* SUDC Subjects whose death was sudden and unexplained after the initial autopsy, and in whom a scene investigation and full autopsy was performed.

Family Members Subjects

* If the SUDC case has DNA viable specimens, family members will be asked if they would also like to participate in the DNA portion. One or both biological parents if willing and able will be considered as a family subject.
* Biological siblings and second degree relatives from age of 0-100 years of age that have had a history or currently have a heart condition and/or neurology condition.

Exclusion Criteria:

SUDC Subjects

* Subjects that are younger than 11months or older than 18 years of age will be excluded as a SUDC case.
* Prospective SUDC cases of apparent suicide, homicide, and accident where the external cause was the obvious and only reason for the death will be excluded from this study.

Family Member Subjects Any siblings or second degree family relatives that did not have a history or current heart or neurology condition will not be able to enroll in the study.

Ages: 11 Months to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1300 participants (400 SUDC subjects and 800 parents, and approximately 100 siblings or symptomatic second degree relatives) over a period of 5 years, including both retrospectively and prospectively ascertained cases.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2014-10-01 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Risks factors leading to sudden unexplained death in childhood (SUDC) collected from PHI | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Orrin Devinsky, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States